CLINICAL TRIAL: NCT01793168
Title: Coordination of Rare Diseases at Sanford
Brief Title: Rare Disease Patient Registry & Natural History Study - Coordination of Rare Diseases at Sanford
Acronym: CoRDS
Status: Recruiting | Type: Observational
Sponsor: Sanford Health (Other)
Collaborators: National Ataxia Foundation (Other); International WAGR Syndrome Association (Unknown); 4p- Support Group (Other); ML4 Foundation (Unknown); Cornelia de Lange Syndrome Foundation (Unknown); Stickler Involved People (Unknown); Kawasaki Disease Foundation (Unknown); Klippel-Feil Syndrome Alliance (Unknown); Klippel-Feil Syndrome Freedom (Unknown); Hyperacusis Research Limited (Unknown); Hypersomnia Foundation (Unknown); Kabuki Syndrome Network (Other); Kleine-Levin Syndrome Foundation (Unknown); Leiomyosarcoma Direct Research Foundation (Unknown); Marinesco-Sjogren Syndrome Support Group - NORD (Other); Mucolipidosis Type IV (ML4) Foundation (Unknown); People with Narcolepsy 4 People with Narcolepsy (PWN4PWN) (Unknown); Soft Bones Incorporated (Unknown); American Multiple Endocrine Neoplasia Support (Unknown); Atypical Hemolytic Uremic Syndrome Foundation (Unknown); All Things Kabuki (Unknown); Wiedemann-Steiner Syndrome Foundation (Unknown); Breast Implant Victim Advocates (Unknown); PROS Foundation (Unknown); American Behcet's Disease Association (Unknown); Alstrom United Kingdom (Unknown); Athymia (Unknown); Curing Retinal Blindness Foundation (Unknown); HSAN1E Society (Unknown); 1p36 Deletion Support and Awareness (Unknown); The Alagille Syndrome Alliance (Unknown); Autoinflammatory Alliance (Unknown); Beyond Batten Disease Foundation (Other); Bohring-Opitz Syndrome Foundation, INC (Unknown); Cockayne Syndrome Network (Share and Care) (Unknown); CRMO Foundation (Unknown); Cure VCP Disease,INC (Unknown); FOD Support (Unknown); Cystinosis Research Foundation (Other); Global DARE Foundation (Unknown); Hypnic Jerk-Sleep Myoclonus Support Group (Unknown); Jansen's Foundation (Unknown); KCNMA1 Channelopathy International Advocacy Foundation (Unknown); Kawasaki Disease Foundation Australia (Unknown); Life with LEMS Foundation (Unknown); Lowe Syndrome Association (Unknown); The Malan Syndrome Foundation (Unknown); Maple Syrup Urine Disease Family Support Group (Unknown); International Association for Muscle Glycogen Storage Disease (IamGSD) (Unknown); Myhre Syndrome Foundation (Unknown); DNM1 Families (Unknown); Nicolaides Baraitser Syndrome (NCBRS) Worldwide Foundation (Unknown); The PBCers Organization (Other); Pitt Hopkins Research Foundation (Other); Recurrent Meningitis Association (Unknown); Recurrent Respiratory Papillomatosis Foundation (Unknown); Remember the Girls (Unknown); Smith-Kingsmore Syndrome Foundation (Unknown); SPG Research Foundation (Unknown); Team Telomere (Unknown); Transient Global Amnesia Project (Unknown); The Charlotte & Gwenyth Gray Foundation (Unknown); The Cute Syndrome Foundation (Unknown); The Maddi Foundation (Unknown); White Sutton Syndrome Foundation (Unknown); Zmynd11 Gene Disorder (Unknown); Cauda Equina Foundation, Inc (Unknown); Tango2 Research Foundation (Unknown); Noah's Hope - Hope4Bridget Foundation (Unknown); Project Sebastian (Unknown); SMC1A Epilepsy Foundation (Unknown); International Foundation for Gastrointestinal Disorders (Unknown); Endosalpingiosis Foundation, Inc (Unknown); International Sacral Agenesis/Caudal Regression Association (ISACRA) (Unknown); Scheuermann's Disease Fund (Unknown); Batten Disease Support and Research Association (Unknown); Kennedy's Disease Association (Unknown); Cure Mito Foundation (Unknown); Warburg Micro Research Foundation (Unknown); Cure Mucolipidosis (Unknown); Riaan Research Initiative (Unknown); CureARS A NJ Nonprofit Corporation (Unknown); CACNA1H Alliance (Unknown); IMBS Alliance (Unknown); SHINE-Syndrome Foundaion (Unknown); Non- Ketotic Hyperglycinemia (NKH) Crusaders (Unknown); Hypertrophic Olivary Degeneration Association (HODA) (Unknown); National Organization for Disorders of the Corpus Callosum (NODCC) (Unknown); Team4Travis (Unknown); Taylor's Tale Foundation (Unknown); Lambert Eaton (LEMS) Family Association (Unknown); BARE Inc (Unknown); STAG1 Gene Foundation (Unknown); Coffin Lowry Syndrome Foundation (Unknown); BLFS Incorporate (Unknown); Aniridia North America (Unknown); Cure Blau Syndrome Foundation (Unknown); ARG1D Foundation (Unknown); CURE HSPB8 Myopathy (Unknown); International Society of Mannosidosis and Related Disorders (Unknown); TBX4Life (Unknown); Cure DHDDS (Unknown); MANDKind Foundation (Unknown); Krishnan Family Foundation (Unknown); SPATA Foundation (Unknown); Acrodysostosis Support and Research (Unknown); ACTA2 Alliance (Unknown); ANA-Aniridia North America (Unknown); CRELD1 Warriors (Unknown); GNB1 Advocacy Group (Unknown); Hope for PDCD Foundation (Unknown); ISMRD - Beta Mannosidosis (Unknown); KBG Syndrome Association (Unknown); The LCC Foundation (Unknown); MLD Foundation (Unknown); MSA United Research Consortium (Unknown); Moyamoya Foundation (Unknown); OPMD Association (Unknown); SKDEAS Foundation (Unknown); The Foundation for Casey's Cure (Unknown); TUBB3 Foundation (Unknown); WWOX Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 03-10-014; Hypersomnia Foundation (Registry Identifier: Hypersomnia Registry); National Ataxia Foundation (Registry Identifier: Ataxia Registry); 4p- Support Group (Registry Identifier: 4p-/Wolfhirschhorn Syndrome Registry); CdLS Foundation (Registry Identifier: Cornelia de Lange Syndrome Registry); Hyperacusis Research Limited (Registry Identifier: Hyperacusis Registry); Kabuki Syndrome Network (Registry Identifier: Kabuki Syndrome Registry); Kawasaki Disease Foundation (Registry Identifier: Kawasaki Disease Registry); Klippel-Feil Syndrome Freedom (Registry Identifier: Klippel-Feil Syndrome Registry); Leiomyosarcoma Direct Research (Registry Identifier: Leiomyosarcoma Registry); MSS Support Group (Registry Identifier: Marinesco-Sjogren Syndrome Registry); ML4 Foundation (Registry Identifier: Mucolipidosis Type IV (ML4) Registry); Stickler Involved People (Registry Identifier: Stickler Syndrome Registry); IWSA (Registry Identifier: WAGR Syndrome Registry); Soft Bones (Registry Identifier: Hypophosphatasia Registry); PWN4PWN (Registry Identifier: Narcolepsy Registry); aHUS (Registry Identifier: aHUS Registry); Klippel-Feil Syndrome Alliance (Registry Identifier: KFS Registry); American MEN Support (Registry Identifier: Mulitiple Endocrine Neoplasia Registry); Kleine-Levin Syndrome (Registry Identifier: Kleine-Levin Syndrome Registry); All Things Kabuki (Registry Identifier: Kabuki Syndrome Registry); WSS Foundation (Registry Identifier: Wiedemann-Steiner Syndrome Registry); BIVA (Registry Identifier: Brest Implant-Associated ALCL Registry); ABDA (Registry Identifier: American Bechet's Disease Association Registry); PROS Foundation (HLH) (Registry Identifier: (HLH) Registry); Alagille Syndrome Association (Registry Identifier: Alagillle Syndrome Registry); Cure VCP Disease, Inc. (Registry Identifier: IBMPFD Registry); Lowe Syndrome Association (Registry Identifier: Lowe Syndrome Registry); Pitt Hopkins (Registry Identifier: Pitt Hopkins Registry); Cure Batten Disease (Registry Identifier: Batten Disease Registry); Hypnic Jerk/Sleep Myoclonus (Registry Identifier: Hypnic Jerk/Sleep Myoclonus Registry); 1p36 DSA (Registry Identifier: 1p36 Deletion Syndrome Registry); Jansen Foundation (Registry Identifier: The Jansen Foundation Registry); Share and Care Network (Registry Identifier: Cockayne Syndrome Registry); CRMO (Registry Identifier: CRMO Registry); The Malan Syndrome Foundation (Registry Identifier: Malan Syndrome Registry); HSAN1E Society (Registry Identifier: HSAN1E Registry); Alstrom United Kingdomg (Registry Identifier: Alstrom United Kingdom Registry); Athymia (Registry Identifier: Athymia Registry); CRB1 Foundation (Registry Identifier: Curing Retinal Blindness Foundation Registry); DNM1 Families (Registry Identifier: DNM1 Mutations Registry); Global DARE Foundation (Registry Identifier: Global DARE Foundation Registry); KCIAF (Registry Identifier: KCNMA1 Channelopathy International Advocacy Foundation Registry); MSUD FSG (Registry Identifier: Maple Syrup Urine Disease Family Support Group Registry); IamGSD (Registry Identifier: International Association for Muscle Glycogen Storage Disease Registry); Myhre Syndrome Foundation (Registry Identifier: Myhre Syndrome Foundation Registry); NCBRS (Registry Identifier: Nicolaides Baraitser Syndrome Worldwide Foundation Registry); PBCers Organization (Registry Identifier: PBCers Organization Registry); Remember the Girls (Registry Identifier: Remember the Girls - X-Linked Carriers Registry); RRPF (Registry Identifier: Recurrent Respiratory Papillomatosis Foundation Registry); SKS Foundation (Registry Identifier: Smith-Kingsmore Syndrome Foundation Registry); SPG15 Research Foundation (Registry Identifier: SPG Research Foundation Registry); Team Telomere (Registry Identifier: Team Telomere Registry); TGA Project (Registry Identifier: Transient Global Amnesia Project Registry); The Cute Syndrome Foundation (Registry Identifier: The Cute Syndrome Foundation Registry); WSS Foundation (Registry Identifier: White Sutton Syndrome Foundation Registry); Zmynd11 Gene Disorder (Registry Identifier: Zmynd11 Gene Disorder Registry); SPG11 and SPG15 (Registry Identifier: The Maddi Foundation Registry); Endosalpingiosis Foundation (Registry Identifier: Endosalpingiosis Foundation, Inc Registry); Cauda Equina Foundation (Registry Identifier: Cauda Equina Foundation, Inc Registry); Tango2 Research Foundation (Registry Identifier: Tango2 Research Foundation Registry); SMC1A Epilepsy (Registry Identifier: SMC1A Epilepsy Foundation Registry); IFFGD (Registry Identifier: International Foundation for Gastrointestinal Disorders); Noah's Hope - Hope4Bridget (Registry Identifier: Noah's Hope - Hope4Bridget Foundation Registry); Project Sebastian (Registry Identifier: Project Sebastian Registry); ISACRA (Registry Identifier: International Sacral Agenesis/Caudal Regression Association (SACRA)); Scheuermann's Disease Fund (Registry Identifier: Scheuermann's Disease Fund Registry); BDSRA (Registry Identifier: Batten Disease Support and Research Association); Kennedy's Disease Assocation (Registry Identifier: Kennedy's Disease Association Registry); Cystinosis Research Foundation (Registry Identifier: Cystinosis Research Foundation Registry); Cure Mito Foundation (Registry Identifier: Cure Mito Foundation Registry); Warburg Micro Research (Registry Identifier: Warburg Micro Research Foundation Registry); Riaan Research Initiative (Registry Identifier: Riaan Research Initiative Registry); Cure Mucolipidosis (Registry Identifier: Cure Mucolipidosis Registry); CACNA1H Alliance (Registry Identifier: CACNA1H Alliance Registry); IMBS Alliance (Registry Identifier: IMBS Alliance Registry); Non-Ketotic Hyperglycinemia (Registry Identifier: NKH Crusaders Registry); Corpus Callosum Disorders (Registry Identifier: NODCC Registry); SHINE Syndrome Foundation (Registry Identifier: SHINE Syndrome Foundation Registry); HODA (Registry Identifier: HODA Registry); Team4Travis (Registry Identifier: Team4Travis Registry); Taylor's Tale Foundation (Registry Identifier: Taylor's Tale Foundation Registry); Lambert Eaton (LEMS) Family (Registry Identifier: (LEMS) Family Association Registry); BARE Inc. (Registry Identifier: BARE Inc. Registry); STAG1 Gene Foundation (Registry Identifier: STAG1 Gene Foundation Registry); Coffin Lowry Syndrome (Registry Identifier: CLS Foundation Registry); BLFS Incorporate (Registry Identifier: BLFS Incorporate Registry); Aniridia North America (Registry Identifier: Aniridia North America Registry); Cure Blau Syndrome Foundation (Registry Identifier: Cure Blau Syndrome Foundation Registry); ARG1D Foundation (Registry Identifier: ARG1D Foundation Registry); CURE HSPB8 Myopathy (Registry Identifier: CURE HSPB8 Myopathy Registry); ISMRD - Beta Mannosidosis (Registry Identifier: ISMRD Registry); TBX4Life (Registry Identifier: TBX4Life Registry); Cure DHDDS (Registry Identifier: Cure DHDDS Registry); MANDKind Foundation (Registry Identifier: MANDKind Foundation Registry); Krishnan Family Foundation (Registry Identifier: Krishnan Family Foundation Registry); SPATA Foundation (Registry Identifier: SPATA Foundation Registry); Acrodysostosis Research (Registry Identifier: 1. Acrodysostosis Support and Research Registry); ACTA2 Alliance (Registry Identifier: ACTA2 Alliance Registry); ANA-Aniridia North America (Registry Identifier: ANA-Aniridia North America Registry); APDS Advocacy Coalition (Registry Identifier: APDS Advocacy Coalition); CRELD1 Warriors (Registry Identifier: CRELD1 Warriors); GNB1 Advocacy Group (Registry Identifier: GNB1 Advocacy Group); Hope for PDCD Foundation (Registry Identifier: Hope for PDCD Foundation); ISMRD - Beta Mannosidosis (Registry Identifier: ISMRD - Beta Mannosidosis); KBG Syndrome Association (Registry Identifier: KBG Syndrome Association Registry); The LCC Foundation (Registry Identifier: The LCC Foundation Registry); MLD Foundation (Registry Identifier: MLD Foundation Registry); MSA United Research (Registry Identifier: MSA United Research Consortium Registry); Moyamoya Foundation (Registry Identifier: Moyamoya Foundation Registry); OPHN1 (Registry Identifier: OPHN1 Registry); OPMD Association (Registry Identifier: OPMD Association Registry); SKDEAS Foundation (Registry Identifier: SKDEAS Foundation Registry); Foundation for Casey's Cure (Registry Identifier: The Foundation for Casey's Cure Registry); TUBB3 Foundation (Registry Identifier: TUBB3 Foundation Registry); WWOX Foundation (Registry Identifier: WWOX Foundation Registry)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Rare Disorders; Undiagnosed Disorders; Disorders of Unknown Prevalence; Cornelia De Lange Syndrome; Prenatal Benign Hypophosphatasia; Perinatal Lethal Hypophosphatasia; Odontohypophosphatasia; Adult Hypophosphatasia; Childhood-onset Hypophosphatasia; Infantile Hypophosphatasia; Hypophosphatasia; Kabuki Syndrome; Bohring-Opitz Syndrome; Narcolepsy Without Cataplexy; Narcolepsy-cataplexy; Hypersomnolence Disorder; Idiopathic Hypersomnia Without Long Sleep Time; Idiopathic Hypersomnia With Long Sleep Time; Idiopathic Hypersomnia; Kleine-Levin Syndrome; Kawasaki Disease; Leiomyosarcoma; Leiomyosarcoma of the Corpus Uteri; Leiomyosarcoma of the Cervix Uteri; Leiomyosarcoma of Small Intestine; Acquired Myasthenia Gravis; Addison Disease; Hyperacusis (Hyperacousis); Juvenile Myasthenia Gravis; Transient Neonatal Myasthenia Gravis; Williams Syndrome; Lyme Disease; Myasthenia Gravis; Marinesco Sjogren Syndrome(Marinesco-Sjogren Syndrome); Isolated Klippel-Feil Syndrome; Frasier Syndrome; Denys-Drash Syndrome; Beckwith-Wiedemann Syndrome; Emanuel Syndrome; Isolated Aniridia; Axenfeld-Rieger Syndrome; Aniridia-intellectual Disability Syndrome; Aniridia - Renal Agenesis - Psychomotor Retardation; Aniridia - Ptosis - Intellectual Disability - Familial Obesity; Aniridia - Cerebellar Ataxia - Intellectual Disability; Aniridia - Absent Patella; Aniridia; Peters Anomaly - Cataract; Peters Anomaly; Potocki-Shaffer Syndrome; Silver-Russell Syndrome Due to Maternal Uniparental Disomy of Chromosome 11; Silver-Russell Syndrome Due to Imprinting Defect of 11p15; Silver-Russell Syndrome Due to 11p15 Microduplication; Syndromic Aniridia; WAGR Syndrome; Wolf-Hirschhorn Syndrome; 4p16.3 Microduplication Syndrome; 4p Deletion Syndrome, Non-Wolf-Hirschhorn Syndrome; Autosomal Recessive Stickler Syndrome; Stickler Syndrome Type 2; Stickler Syndrome Type 1; Stickler Syndrome; Mucolipidosis Type 4; X-linked Spinocerebellar Ataxia Type 4; X-linked Spinocerebellar Ataxia Type 3; X-linked Intellectual Disability - Ataxia - Apraxia; X-linked Progressive Cerebellar Ataxia; X-linked Non Progressive Cerebellar Ataxia; X-linked Cerebellar Ataxia; Vitamin B12 Deficiency Ataxia; Toxic Exposure Ataxia; Unclassified Autosomal Dominant Spinocerebellar Ataxia; Thyroid Antibody Ataxia; Sporadic Adult-onset Ataxia of Unknown Etiology; Spinocerebellar Ataxia With Oculomotor Anomaly; Spinocerebellar Ataxia With Epilepsy; Spinocerebellar Ataxia With Axonal Neuropathy Type 2; Spinocerebellar Ataxia Type 8; Spinocerebellar Ataxia Type 7; Spinocerebellar Ataxia Type 6; Spinocerebellar Ataxia Type 5; Spinocerebellar Ataxia Type 4; Spinocerebellar Ataxia Type 37; Spinocerebellar Ataxia Type 36; Spinocerebellar Ataxia Type 35; Spinocerebellar Ataxia Type 34; Spinocerebellar Ataxia Type 32; Spinocerebellar Ataxia Type 31; Spinocerebellar Ataxia Type 30; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 29; Spinocerebellar Ataxia Type 28; Spinocerebellar Ataxia Type 27; Spinocerebellar Ataxia Type 26; Spinocerebellar Ataxia Type 25; Spinocerebellar Ataxia Type 23; Spinocerebellar Ataxia Type 22; Spinocerebellar Ataxia Type 21; Spinocerebellar Ataxia Type 20; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 19/22; Spinocerebellar Ataxia Type 18; Spinocerebellar Ataxia Type 17; Spinocerebellar Ataxia Type 16; Spinocerebellar Ataxia Type 15/16; Spinocerebellar Ataxia Type 14; Spinocerebellar Ataxia Type 13; Spinocerebellar Ataxia Type 12; Spinocerebellar Ataxia Type 11; Spinocerebellar Ataxia Type 10; Spinocerebellar Ataxia Type 1 With Axonal Neuropathy; Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia - Unknown; Spinocerebellar Ataxia - Dysmorphism; Non Progressive Epilepsy and/or Ataxia With Myoclonus as a Major Feature; Spasticity-ataxia-gait Anomalies Syndrome; Spastic Ataxia With Congenital Miosis; Spastic Ataxia - Corneal Dystrophy; Spastic Ataxia; Rare Hereditary Ataxia; Rare Ataxia; Recessive Mitochondrial Ataxia Syndrome; Progressive Epilepsy and/or Ataxia With Myoclonus as a Major Feature; Posterior Column Ataxia - Retinitis Pigmentosa; Post-Stroke Ataxia; Post-Head Injury Ataxia; Post Vaccination Ataxia; Polyneuropathy - Hearing Loss - Ataxia - Retinitis Pigmentosa - Cataract; Muscular Atrophy - Ataxia - Retinitis Pigmentosa - Diabetes Mellitus; Non-hereditary Degenerative Ataxia; Paroxysmal Dystonic Choreathetosis With Episodic Ataxia and Spasticity; Olivopontocerebellar Atrophy - Deafness; NARP Syndrome; Myoclonus - Cerebellar Ataxia - Deafness; Multiple System Atrophy, Parkinsonian Type; Multiple System Atrophy, Cerebellar Type; Multiple System Atrophy; Maternally-inherited Leigh Syndrome; Machado-Joseph Disease Type 3; Machado-Joseph Disease Type 2; Machado-Joseph Disease Type 1; Leigh Syndrome; Late-onset Ataxia With Dementia; Infection or Post Infection Ataxia; GAD Ataxia; Hereditary Episodic Ataxia; Gliadin/Gluten Ataxia; Friedreich Ataxia; Fragile X-associated Tremor/Ataxia Syndrome; Familial Paroxysmal Ataxia; Exposure to Medications Ataxia; Episodic Ataxia With Slurred Speech; Episodic Ataxia Unknown Type; Episodic Ataxia Type 7; Episodic Ataxia Type 6; Episodic Ataxia Type 5; Episodic Ataxia Type 4; Episodic Ataxia Type 3; Episodic Ataxia Type 1; Epilepsy and/or Ataxia With Myoclonus as Major Feature; Early-onset Spastic Ataxia-neuropathy Syndrome; Early-onset Progressive Neurodegeneration - Blindness - Ataxia - Spasticity; Early-onset Cerebellar Ataxia With Retained Tendon Reflexes; Early-onset Ataxia With Dementia; Childhood-onset Autosomal Recessive Slowly Progressive Spinocerebellar Ataxia; Dilated Cardiomyopathy With Ataxia; Cataract - Ataxia - Deafness; Cerebellar Ataxia, Cayman Type; Cerebellar Ataxia With Peripheral Neuropathy; Cerebellar Ataxia - Hypogonadism; Cerebellar Ataxia - Ectodermal Dysplasia; Cerebellar Ataxia - Areflexia - Pes Cavus - Optic Atrophy - Sensorineural Hearing Loss; Brain Tumor Ataxia; Brachydactyly - Nystagmus - Cerebellar Ataxia; Benign Paroxysmal Tonic Upgaze of Childhood With Ataxia; Autosomal Recessive Syndromic Cerebellar Ataxia; Autosomal Recessive Spastic Ataxia With Leukoencephalopathy; Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay; Autosomal Recessive Spastic Ataxia - Optic Atrophy - Dysarthria; Autosomal Recessive Spastic Ataxia; Autosomal Recessive Metabolic Cerebellar Ataxia; Autosomal Dominant Spinocerebellar Ataxia Due to Repeat Expansions That do Not Encode Polyglutamine; Autosomal Recessive Ataxia, Beauce Type; Autosomal Recessive Ataxia Due to Ubiquinone Deficiency; Autosomal Recessive Ataxia Due to PEX10 Deficiency; Autosomal Recessive Degenerative and Progressive Cerebellar Ataxia; Autosomal Recessive Congenital Cerebellar Ataxia Due to MGLUR1 Deficiency; Autosomal Recessive Congenital Cerebellar Ataxia Due to GRID2 Deficiency; Autosomal Recessive Congenital Cerebellar Ataxia; Autosomal Recessive Cerebellar Ataxia-pyramidal Signs-nystagmus-oculomotor Apraxia Syndrome; Autosomal Recessive Cerebellar Ataxia-epilepsy-intellectual Disability Syndrome Due to WWOX Deficiency; Autosomal Recessive Cerebellar Ataxia-epilepsy-intellectual Disability Syndrome Due to TUD Deficiency; Autosomal Recessive Cerebellar Ataxia-epilepsy-intellectual Disability Syndrome Due to KIAA0226 Deficiency; Autosomal Recessive Cerebellar Ataxia-epilepsy-intellectual Disability Syndrome; Autosomal Recessive Cerebellar Ataxia With Late-onset Spasticity; Autosomal Recessive Cerebellar Ataxia Due to STUB1 Deficiency; Autosomal Recessive Cerebellar Ataxia Due to a DNA Repair Defect; Autosomal Recessive Cerebellar Ataxia - Saccadic Intrusion; Autosomal Recessive Cerebellar Ataxia - Psychomotor Retardation; Autosomal Recessive Cerebellar Ataxia - Blindness - Deafness; Autosomal Recessive Cerebellar Ataxia; Autosomal Dominant Spinocerebellar Ataxia Due to a Polyglutamine Anomaly; Autosomal Dominant Spinocerebellar Ataxia Due to a Point Mutation; Autosomal Dominant Spinocerebellar Ataxia Due to a Channelopathy; Autosomal Dominant Spastic Ataxia Type 1; Autosomal Dominant Spastic Ataxia; Autosomal Dominant Optic Atrophy; Ataxia-telangiectasia Variant; Ataxia-telangiectasia; Autosomal Dominant Cerebellar Ataxia, Deafness and Narcolepsy; Autosomal Dominant Cerebellar Ataxia Type 4; Autosomal Dominant Cerebellar Ataxia Type 3; Autosomal Dominant Cerebellar Ataxia Type 2; Autosomal Dominant Cerebellar Ataxia Type 1; Autosomal Dominant Cerebellar Ataxia; Ataxia-telangiectasia-like Disorder; Ataxia With Vitamin E Deficiency; Ataxia With Dementia; Ataxia - Oculomotor Apraxia Type 1; Ataxia - Other; Ataxia - Genetic Diagnosis - Unknown; Acquired Ataxia; Adult-onset Autosomal Recessive Cerebellar Ataxia; Alcohol Related Ataxia; Multiple Endocrine Neoplasia; Multiple Endocrine Neoplasia Type II; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2; Multiple Endocrine Neoplasia, Type IV; Multiple Endocrine Neoplasia, Type 3; Multiple Endocrine Neoplasia (MEN) Syndrome; Multiple Endocrine Neoplasia Type 2B; Multiple Endocrine Neoplasia Type 2A; Atypical Hemolytic Uremic Syndrome; Atypical HUS; Wiedemann-Steiner Syndrome; Breast Implant-Associated Anaplastic Large Cell Lymphoma; Autoimmune/Inflammatory Syndrome Induced by Adjuvants (ASIA); Hemophagocytic Lymphohistiocytosis; Behcet's Disease; Alagille Syndrome; Inclusion Body Myopathy With Early-onset Paget Disease and Frontotemporal Dementia (IBMPFD); Lowe Syndrome; Pitt Hopkins Syndrome; 1p36 Deletion Syndrome; Jansen Type Metaphyseal Chondrodysplasia; Cockayne Syndrome; Chronic Recurrent Multifocal Osteomyelitis; CRMO; Malan Syndrome; Hereditary Sensory and Autonomic Neuropathy Type Ie; VCP Disease; Hypnic Jerking; Sleep Myoclonus; Mollaret Meningitis; Recurrent Viral Meningitis; CRB1; Leber Congenital Amaurosis; Retinitis Pigmentosa; Rare Retinal Disorder; KCNMA1-Channelopathy; Primary Biliary Cirrhosis; ZMYND11; Transient Global Amnesia; Glycogen Storage Disease; Alstrom Syndrome; White Sutton Syndrome; DNM1; EIEE31; Myhre Syndrome; Recurrent Respiratory Papillomatosis; Laryngeal Papillomatosis; Tracheal Papillomatosis; Refsum Disease; Nicolaides Baraitser Syndrome; Leukodystrophy; Tango2; Cauda Equina Syndrome; Rare Gastrointestinal Disorders; Achalasia-Addisonian Syndrome; Achalasia Cardia; Achalasia Icrocephaly Syndrome; Anal Fistula; Congenital Sucrase-Isomaltase Deficiency; Eosinophilic Gastroenteritis; Idiopathic Gastroparesis; Hirschsprung Disease; Rare Inflammatory Bowel Disease; Intestinal Pseudo-Obstruction; Scleroderma; Short Bowel Syndrome; Sacral Agenesis; Sacral Agenesis Syndrome; Caudal Regression; Scheuermann Disease; SMC1A Truncated Mutations (Causing Loss of Gene Function); Cystinosis; Juvenile Nephropathic Cystinosis; Nephropathic Cystinosis; Kennedy Disease; Spinal Bulbar Muscular Atrophy; Warburg Micro Syndrome; Mucolipidoses; Mitochondrial Diseases; Mitochondrial Aminoacyl-tRNA Synthetases; Mt-aaRS Disorders; Hypertrophic Olivary Degeneration; Non-Ketotic Hyperglycinemia; Fish Odor Syndrome; Halitosis; Isolated Congenital Asplenia; Lambert Eaton (LEMS); Biliary Atresia; STAG1 Gene Mutation; Coffin Lowry Syndrome; Borjeson-Forssman-Lehman Syndrome; Blau Syndrome; Arginase 1 Deficiency; HSPB8 Myopathy; Beta-Mannosidosis; TBX4 Syndrome; DHDDS Gene Mutations; MAND-MBD5-Associated Neurodevelopmental Disorder; Constitutional Mismatch Repair Deficiency (CMMRD); SPATA5 Disorder; SPATA5L1 Related Disorder; Acrodysostosis; Multi-systematic Smooth Muscle Dysfunction Syndrome; CRELD1 (Cysteine Rich With EGF Like Domains 1); GNB1 Syndrome; Pyruvate Dehydrogenase Complex Deficiency Disease; Beta Mannosidosis; Kbg Syndrome; Labrune Syndrome; Metachromatic Leukodystrophy (MLD); Moyamoya Disease; OPHN1 Syndrome; Oculopharyngeal Muscular Dystrophy (OPMD); TUBB3 Mutation; WOREE (WWOX-related Epileptic Encephalopathy; SCAR12; Skraban-Deardorff Syndrome; Hereditary Myopathy With Early Respiratory Failure
Keywords: Rare Diseases; Neglected Diseases; Orphan Diseases; Rare Disease Research; Registries; WAGR Syndrome; Ataxia; Cornelia de Lange Syndrome; Stickler Syndrome; Ataxia Telangiectasia; Kawasaki Disease; Batten Disease; Mucolipidosis IV; Klippel-Feil Syndrome; Multiple Endocrine Neoplasia; Atypical Hemolytic Uremic Syndrome; Undiagnosed; Uncommon Disease; Kabuki Syndrome; Hypersomnia; Hyperacusis; Kleine-Levin Syndrome; Marinesco-Sjogren Syndrome; Leiomyosarcoma; 4p-/Wolf-Hirschhorn Syndrome; Hypophosphatasia; Narcolepsy; Wiedermann-Steiner Syndrome; Breast Implant-Associated Anaplastic Large Cell Lymphoma; Autoimmune/inflammatory Syndrome Induced by Adjuvants (ASIA); Hemophagocytic Lymphohistiocytosis (HLH); Behcet's Disease; Alagille Syndrome; Inclusion body myopathy with early-onset Paget disease and frontotemporal dementia (IBMPFD); Lowe Syndrome; Pitt Hopkins Syndrome; 1p36 deletion syndrome; Jansen metaphyseal chondrodysplasia; Cockayne Syndrome; Chronic recurrent multifocal osteomyelitis (CRMO); Malan syndrome; Hereditary Sensory and Autonomic Neuropathy; Cystinosis; Juvenile nephropathic cystinosis; Nephropathic infantile cystinosis; Ocular cystinosis; Kennedy disease; Spinal Bulbar Muscular Atrophy (SBMA); SMC1A Truncated Mutations (causing loss of gene function); Leigh syndrome; Warburg Micro Syndrome; Mucolipidosis; Mitochondrial aminoacyl-tRNA synthetases (Mt-aaRS Disorders); Shine Syndrome; Hypertrophic Olivary Degeneration; Non-Ketotic Hyperglycinemia; Intestinal Bromhidrosis Syndrome; Fish odor syndrome; Autosomal recessive extra oral halitosis; CACNA1H mutation; Dimethylglycine dehydrogenase deficiency
MeSH Terms: conditions — De Lange Syndrome; Hypophosphatasia, Perinatal Lethal; Odontohypophosphatasia; Hypophosphatasia, Adult; Hypophosphatasia, Childhood; Hypophosphatasia; Kabuki syndrome; Bohring syndrome; Narcolepsy; Disorders of Excessive Somnolence; Idiopathic Hypersomnia; Kleine-Levin Syndrome; Mucocutaneous Lymph Node Syndrome; Leiomyosarcoma; Addison Disease; Hyperacusis; Myasthenia Gravis, Neonatal; Williams Syndrome; Lyme Disease; Myasthenia Gravis; Spinocerebellar Degenerations; Frasier Syndrome; Denys-Drash Syndrome; Beckwith-Wiedemann Syndrome; Emanuel syndrome; Axenfeld-Rieger syndrome; Aniridia, Partial, with Unilateral Renal Agenesis and Psychomotor Retardation; Aniridia and Absent Patella; Aniridia; Peters anomaly; Potocki-Shaffer syndrome; WAGR Syndrome; Wolf-Hirschhorn Syndrome; Stickler syndrome, type 2; Stickler syndrome, type 1; Mucolipidoses; Spinocerebellar ataxia, X-linked, 4; Spinocerebellar ataxia, X-linked, 3; Spinocerebellar Ataxia with Epilepsy; Spinocerebellar ataxia, autosomal recessive 1; Spinocerebellar ataxia 8; Spinocerebellar Ataxias; Erythrokeratodermia with ataxia; Spinocerebellar Ataxia 31; Spinocerebellar ataxia 30; Machado-Joseph Disease; Spinocerebellar Ataxia 15; Spinocerebellar ataxia 28; Spinocerebellar ataxia 27; Spinocerebellar ataxia 26; Spinocerebellar ataxia 25; Spinocerebellar ataxia 23; Spinocerebellar ataxia 21; Spinocerebellar ataxia 20; Sensorimotor neuropathy with ataxia, autosomal dominant; Olivopontocerebellar Atrophy V; Spinocerebellar ataxia 14; Spinocerebellar ataxia 13; Spinocerebellar Ataxia 12; Spinocerebellar Ataxia 11; Spinocerebellar Ataxia 10; Ataxia, Spastic, with Congenital Miosis; Spastic Ataxia; Ataxia Neuropathy Spectrum; Polyneuropathy, Hearing Loss, Ataxia, Retinitis Pigmentosa, And Cataract; Muscular Atrophy, Ataxia, Retinitis Pigmentosa, and Diabetes Mellitus; Muscle Spasticity; Neuropathy ataxia and retinitis pigmentosa; Myoclonus, Cerebellar Ataxia, and Deafness; Multiple System Atrophy; Maternally Inherited Leigh Syndrome; Leigh Disease; Infections; Friedreich Ataxia; Fragile X Tremor Ataxia Syndrome; Episodic Ataxia, Type 2; Episodic Ataxia, Type 7; Episodic Ataxia, Type 6; Episodic Ataxia, Type 5; Episodic Ataxia, Type 4; Episodic Ataxia, Type 3; Episodic Ataxia, Type 1; Harding ataxia; Spinocerebellar Ataxia, Autosomal Recessive 7; 3-Methylglutaconic Aciduria, Type V; Cataract ataxia deafness; Cerebellar Ataxia, Cayman Type; Cerebellar Ataxia and Hypogonadotropic Hypogonadism; Cerebellar ataxia ectodermal dysplasia; CAPOS syndrome; Brachydactyly-Nystagmus-Cerebellar Ataxia; Paroxysmal Tonic Upgaze, Benign Childhood, With Ataxia; Ataxia, Spastic, 3, Autosomal Recessive; Spastic ataxia Charlevoix-Saguenay type; Spinocerebellar Ataxia, Autosomal Recessive 8; Spinocerebellar ataxia, autosomal recessive 3; Optic Atrophy, Autosomal Dominant; Ataxia-Telangiectasia Variant; Ataxia Telangiectasia; Deafness; Ataxia Telangiectasia Like Disorder; Ataxia with vitamin E deficiency; Early-onset ataxia with oculomotor apraxia and hypoalbuminemia; Multiple Endocrine Neoplasia; Multiple Endocrine Neoplasia Type 2a; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia, Type IV; Multiple Endocrine Neoplasia Type 2b; Syndrome; Atypical Hemolytic Uremic Syndrome; Growth Deficiency and Mental Retardation with Facial Dysmorphism; Lymphohistiocytosis, Hemophagocytic; Alagille Syndrome; Frontotemporal Dementia; Inclusion Body Myopathy With Early-Onset Paget Disease And Frontotemporal Dementia; Oculocerebrorenal Syndrome; Pitt-Hopkins syndrome; Chromosome 1p36 Deletion Syndrome; Jansen type metaphyseal chondrodysplasia; Cockayne Syndrome; Chronic recurrent multifocal osteomyelitis; Hereditary Sensory and Autonomic Neuropathy Type Ie; Myoclonus; Meningitis, Viral; Leber Congenital Amaurosis; Retinitis Pigmentosa; Liver Cirrhosis, Biliary; Amnesia, Transient Global; Glycogen Storage Disease; Alstrom Syndrome; Growth mental deficiency syndrome of Myhre; Recurrent respiratory papillomatosis; Laryngeal papillomatosis; Refsum Disease; Nicolaides Baraitser syndrome; Cauda Equina Syndrome; Achalasia Addisonianism Alacrimia syndrome; Esophageal Achalasia; Rectal Fistula; Sucrase-isomaltase deficiency, congenital; Eosinophilic enteropathy; Hirschsprung Disease; Intestinal Pseudo-Obstruction; Scleroderma, Diffuse; Short Bowel Syndrome; Sacral defect and anterior sacral meningocele; Sacral Agenesis Syndrome; Scheuermann Disease; Cystinosis; Cystinosis, Late-Onset Juvenile or Adolescent Nephropathic Type; Bulbo-Spinal Atrophy, X-Linked; Warburg Sjo Fledelius syndrome; Mitochondrial Diseases; Olivary Degeneration; Hyperglycinemia, Nonketotic; Trimethylaminuria; Halitosis; Lambert-Eaton Myasthenic Syndrome; Biliary Atresia; Coffin-Lowry Syndrome; Blau syndrome; Hyperargininemia; beta-Mannosidosis; Turcot syndrome; Acrodysostosis; Pyruvate Dehydrogenase Complex Deficiency Disease; KBG syndrome; Leukoencephalopathy Brain Calcifications and Cysts; Leukodystrophy, Metachromatic; Moyamoya Disease; Muscular Dystrophy, Oculopharyngeal; Hereditary Myopathy with Early Respiratory Failure; Rare Diseases; Neglected Diseases; Ataxia; Neuronal Ceroid-Lipofuscinoses; Klippel-Feil Syndrome; Hereditary Sensory and Autonomic Neuropathies; Cystinosis, Infantile Nephropathic; Dimethylglycine Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: None Retained — Biospecimen collection capability anticipated in 2014.
Oversight: Data Monitoring Committee: No

SUMMARY:
CoRDS, or the Coordination of Rare Diseases at Sanford, is based at Sanford Research in Sioux Falls, South Dakota. It provides researchers with a centralized, international patient registry for all rare diseases. This program allows patients and researchers to connect as easily as possible to help advance treatments and cures for rare diseases. The CoRDS team works with patient advocacy groups, individuals and researchers to help in the advancement of research in over 7,000 rare diseases. The registry is free for patients to enroll and researchers to access. Visit sanfordresearch.org/CoRDS to enroll.

DETAILED DESCRIPTION:
CoRDS collects contact, sociodemographic and health information about participants. This information is entered into CoRDS and linked to a unique coded identifier. Below are some examples of information requested on the Questionnaire that will be entered into CoRDS:

* Contact information: Name, Mailing Address, Phone Number, Email Address
* Sociodemographic information: Date of Birth, Place of Birth, Sex, Gender, Ethnicity
* Health information: Family History, Information related to Diagnosis

De-identified information in CoRDS will be made available to researchers, if they have obtained approval for their research project from (1) the Institutional Review Board (IRB) at the researcher's institution and (2) a panel of experts.

A subset of de-identified information collected from each profile may be shared with certain other databases. This is done in order to help improve understanding of rare diseases, to avoid the duplication of efforts and to collaborate with existing research efforts with organizations dedicated to rare diseases.

Participants may elect to have their information shared with patient advocacy groups (PAGs) representing individuals with rare or uncommon diseases who have partnered with CoRDS. The PAG will sign an agreement stating that they will not use the information for Research purposes. CoRDS personnel will not be held responsible for the use of information by the PAG.

The CoRDS Registry will not be paid by Researchers, Other Patient Registries or Patient Advocacy Groups (PAGs) for access to information in CoRDS.

If a parent/LAR consents on behalf of a minor, CoRDS will contact the participant when he or she reaches the age of 18 in order to obtain consent. If this consent is not obtained in a timely manner, the participant will be withdrawn from CoRDS.

CoRDS contacts participants annually to confirm continued interest in participation in CoRDS, and to request that participants update the information they have provided.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare disease, a disease of unknown prevalence, undiagnosed or an unaffected carrier of a rare/uncommon disease

Exclusion Criteria:

* Diagnosis of a disease which is not rare

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unaffected carriers, undiagnosed and those with a rare disease or rare condition.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2010-07 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
To accelerate research into rare disorders by connecting individuals who are interested in research and who have been diagnosed with a rare disorder (or a disorder of unknown prevalence, or who are undiagnosed) with researchers who study rare diseases. | 100 years

CONTACTS AND LOCATIONS:
Locations (2):
- Sanford Health, Sioux Falls, South Dakota, United States
- Online Patient Enrollment System, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data is shared with contracted patient advocacy groups for non-research purposes. Parties interested in accessing data are welcome to apply (cost-free) at http://www.sanfordresearch.org/cords/researchers/.

REFERENCES:
- See also: CoRDS homepage — http://www.sanfordresearch.org/SpecialPrograms/cords/
- See also: CoRDS Screening Form — https://cordsconnect.sanfordresearch.org/BayaPES/sf/screeningForm?id=SFSFL#
- See also: CoRDS Participant Login — https://cordsconnect.sanfordresearch.org/BayaPES/pp/participantLogin#